CLINICAL TRIAL: NCT05101031
Title: Evaluation of Fluid Volume in Patients With Refractory Hypotension (Fresh-ER)
Acronym: Fresh-ER
Status: Completed | Type: Observational
Sponsor: Ivor Douglas (Other)
Collaborators: Oregon Health and Science University (Other); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor-Investigator, Ivor Douglas, Chief of Pulmonary and Medical Critical Care, Denver Health and Hospital Authority
Organization: Denver Health and Hospital Authority (Other)
Other Study IDs: 20-2845
Record Dates: First submitted 2021-06-22; First posted 2021-10-29 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Undifferentated Shock
Keywords: Resuscitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Denver Health Medical Center: SV machine will be attached if hypotensive and in the emergency department
  Interventions: Device: Starling SV

INTERVENTIONS:
Device: Starling SV — The Starling SV will monitor the change in hemodynamic variables (i.e. CO, SV, HR, SV) as assessed during the initial fluid resuscitation in individuals with hypotension related to infection.

SUMMARY:
The objective of the study is to observe the change in hemodynamic variables (i.e. CO, SV, HR, SV) as assessed during rapid fluid bolus.

DETAILED DESCRIPTION:
The Noninvasive Starling SV (Baxter Healthcare) is a portable, non-invasive, cardiac output detector system. The Starling SV system measures the cardiac output by employing electrical bioreactance. Bioreactance is a measure of the electrical characteristics of a volume of tissue and fluid. In the case of cardiac output measurements, the relevant tissue includes the heart and the immediate surrounding volume of the thorax. The relevant fluid is blood.

The objective of the study is observe the change in hemodynamic variables (i.e. CO, SV, HR, SV) as assessed during the initial resuscitation of 30 ml/kg of fluid, to evaluate the feasibility of performing a larger prospective RCT of SV-guided resuscitation in patients who undergo a dynamic assessment of fluid responsiveness to help guide fluid administration.

This study is a prospective feasibility study. Patients will be evaluated by the Emergency Room team for Inclusion/Exclusion criteria. If the patient is found to fit the study inclusion and exclusion criteria, then the fully non-invasive Starling monitor will be applied to the patient and the patient's hemodynamic data will be prospectively collected during the initial fluid resuscitation.

ELIGIBILITY:
Inclusion Criteria:

Primary Criteria

1. MAP <65
2. SBP <90 or BP rapidly trending lower

   Secondary Criteria
3. Low urine output Acute change in urine output less than 50ml/4 hours
4. Persistent hyperlactatemia
5. A new vasopressor started
6. Acute change in HR less than 50 or greater than 120
7. New onset chest pain or chest pain different then admission assessment
8. Acute bleeding
9. Fever > 39 degrees
10. Significant change in mental status: confusion, agitation, delirium, etc.
11. Unexplained lethargy
12. CRT >2 seconds -

Exclusion Criteria:

1. Primary diagnosis of: acute cerebral vascular event, acute coronary syndrome, acute pulmonary edema, status asthmatics, major cardiac arrhythmia, drug overdose, or injury from burn or trauma
2. Known aortic insufficiency, or aortic abnormalities
3. Requires immediate surgery
4. Advanced directives restricting implementation of the resuscitation protocol
5. Known intraventricular heart defect, such as VSD or ASD
6. Prisoner
7. Pregnancy
8. Age <18
9. Known allergy to sensor material or gel
10. Suspected intra-abdominal hypertension
11. Inability to obtain IV access
12. Patient should be excluded based on the opinion of the Clinician/Investigator
13. Patient has an unstable airway

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be drawn from all patients who undergo present to the Emergency Room with symptoms of suspected or confirmed septic shock, and who are identified to receive a 30cc/kg fluid bolus of resuscitation fluid as part of treatment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2022-12-17 (Actual); Study Completion 2022-12-17 (Actual)

PRIMARY OUTCOMES:
Stroke Volume Change | During fluid bolus
  Change in stroke volume following the administration of each 500 cc fluid bolus.

SECONDARY OUTCOMES:
Stroke Volume Difference | during fluid bolus
  Concordance between change in stroke volume compared between fluid bolus and other usual care assessments of effective circulating volume
Fluid Input and Output | 72 hours
  Fluid balance inclusive of all parenteral fluids and all output
LOS in ICU | Up to 180 days from ICU admission
  Length of ICU stay (days) until subject is medically ready for discharge
Mechanical ventilation | 28 days
  Requirement for mechanical ventilation during hospitalization
Vasopressor Use | 28 days
  Requirement for vasopressor use during hospitalization
Serum Creatinine Levels | 28 days
  Changes in serum creatinine levels from baseline
Renal Replacement Therapy | 28 days
  Requirement for renal replacement therapy (RRT)
MACE | 28 days
  Incidence of Major Adverse Cardiac Event (MACE)
Adverse Events | 28 days
  Incident of Adverse Events
Mortality | 28 days
  Inhospital Mortality rate
Discharge Location | Up to 180 days from hospital admission
  Discharge location after hospitalization
Fluid Input and Output in ICU | 28 days
  Mean difference in fluid balance at ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Ivor Douglas, MD, Principal Investigator — Denver Health Medical Center
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

REFERENCES:
- [Background] Monnet X, Teboul JL. Passive leg raising. Intensive Care Med. 2008 Apr;34(4):659-63. doi: 10.1007/s00134-008-0994-y. Epub 2008 Jan 23. PMID 18214429
- [Result] Marik PE, Cavallazzi R. Does the central venous pressure predict fluid responsiveness? An updated meta-analysis and a plea for some common sense. Crit Care Med. 2013 Jul;41(7):1774-81. doi: 10.1097/CCM.0b013e31828a25fd. PMID 23774337
- [Result] Michard F, Teboul JL. Predicting fluid responsiveness in ICU patients: a critical analysis of the evidence. Chest. 2002 Jun;121(6):2000-8. doi: 10.1378/chest.121.6.2000. PMID 12065368
- [Result] Kelm DJ, Perrin JT, Cartin-Ceba R, Gajic O, Schenck L, Kennedy CC. Fluid overload in patients with severe sepsis and septic shock treated with early goal-directed therapy is associated with increased acute need for fluid-related medical interventions and hospital death. Shock. 2015 Jan;43(1):68-73. doi: 10.1097/SHK.0000000000000268. PMID 25247784
- [Result] Boyd JH, Forbes J, Nakada TA, Walley KR, Russell JA. Fluid resuscitation in septic shock: a positive fluid balance and elevated central venous pressure are associated with increased mortality. Crit Care Med. 2011 Feb;39(2):259-65. doi: 10.1097/CCM.0b013e3181feeb15. PMID 20975548
- [Result] Vincent et al. Sepsis in European ICU: Results of the SOAP study. British Journal of Anesthesia 2006; 113: 740-747.